CLINICAL TRIAL: NCT07348133
Title: An Open-Label, Randomized, Three-Period, Six-Sequence Phase I Study to Evaluate the Effect of Food on the Pharmacokinetics of HMPL-523 Acetate Tablets in Healthy Participants
Brief Title: Study of Food Effect on Pharmacokinetics of HMPL-523 Acetate Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-523-00CH2
Record Dates: First submitted 2025-11-26; First posted 2026-01-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: HMPL-523

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, randomized, three-period, six-sequence study. There are 3 cycles of dosing, and participants will be randomized to 1 of the 6 dosing sequences (ABC, ACB, BAC, BCA, CAB, or CBA).
  The 3 cycles of each sequence consist of 3 dietary conditions, i.e., fasting (A), standard high-fat breakfast (B), and standard low-fat breakfast (C). Participants will receive a single oral dose of HMPL-523 acetate tablets 300 mg on Day 1 of each cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ABC (Experimental): The 3 cycles of each sequence consist of 3 dietary conditions, i.e., fasting (A), standard high-fat breakfast (B), and standard low-fat breakfast (C). Participants will receive a single oral dose of HMPL-523 acetate tablets 300 mg on Day 1 of each cycle.
  Interventions: Drug: HMPL-523
- ACB (Experimental): The 3 cycles of each sequence consist of 3 dietary conditions, i.e., fasting (A), standard high-fat breakfast (B), and standard low-fat breakfast (C). Participants will receive a single oral dose of HMPL-523 acetate tablets 300 mg on Day 1 of each cycle.
  Interventions: Drug: HMPL-523
- BAC (Experimental): The 3 cycles of each sequence consist of 3 dietary conditions, i.e., fasting (A), standard high-fat breakfast (B), and standard low-fat breakfast (C). Participants will receive a single oral dose of HMPL-523 acetate tablets 300 mg on Day 1 of each cycle.
  Interventions: Drug: HMPL-523
- BCA (Experimental): The 3 cycles of each sequence consist of 3 dietary conditions, i.e., fasting (A), standard high-fat breakfast (B), and standard low-fat breakfast (C). Participants will receive a single oral dose of HMPL-523 acetate tablets 300 mg on Day 1 of each cycle.
  Interventions: Drug: HMPL-523
- CAB (Experimental): The 3 cycles of each sequence consist of 3 dietary conditions, i.e., fasting (A), standard high-fat breakfast (B), and standard low-fat breakfast (C). Participants will receive a single oral dose of HMPL-523 acetate tablets 300 mg on Day 1 of each cycle.
  Interventions: Drug: HMPL-523
- CBA (Experimental): The 3 cycles of each sequence consist of 3 dietary conditions, i.e., fasting (A), standard high-fat breakfast (B), and standard low-fat breakfast (C). Participants will receive a single oral dose of HMPL-523 acetate tablets 300 mg on Day 1 of each cycle.
  Interventions: Drug: HMPL-523

INTERVENTIONS:
Drug: HMPL-523 — The 3 cycles of each sequence consist of 3 dietary conditions, i.e., fasting (A), standard high-fat breakfast (B), and standard low-fat breakfast (C). Participants will receive a single oral dose of HMPL-523 acetate tablets 300 mg on Day 1 of each cycle.

SUMMARY:
This is a single-center, open-label, randomized, three-period, six-sequence study to evaluate the effect of food (high-fat and low-fat) on the PK of HMPL-523. In this study, 18 healthy Chinese participants are planned to be enrolled, randomized in a ratio of 1:1:1:1:1:1 to one of 6 dosing sequences (see dosing sequence table for details), and administered once per cycle for 3 cycles, with a washout period of at least 7 days. The study consists of a screening/baseline period, a dosing period (three cycles), and a follow-up period.

DETAILED DESCRIPTION:
Screening Period/Baseline Period The trial participants will sign a written informed consent form on a voluntary basis prior to screening. Screening period/baseline period assessment will be completed within 14 days prior to the first dose. At screening/baseline, demographic data, medical history, medication history, allergy history, blood donation history, and participation in clinical trials should be collected, and physical examination, vital sign measurements, 12-lead ECG, infection markers, laboratory tests, pregnancy test , and chest X-ray will be performed.

Trial participants who pass the preliminary screening will be admitted to the study site 3 days prior to the first dose (i.e., 3 days prior to medication of Cycle 1), vital signs examination, urine drug abuse screening, alcohol breath screening will be performed on the day of admission, recent dietary and medication use will be inquired, and pregnancy test will be conducted (only for women of childbearing potential. If the screening examinations and baseline examinations will be conducted on the same day, they can be done once), and the inclusion and exclusion criteria will be further checked.

Only serious adverse events will be collected during screening/baseline period. Dosing Period (3 cycles) The day before the first administration, trial participants passing the screening will be given a randomization number according to the randomization scheme, and assigned to one of 6 dosing sequences in a ratio of 1:1:1:1:1:1. The dosing sequences include ABC, ACB, BAC, BCA, CAB and CBA, and the three dietary conditions are fasting (A), standard high-fat breakfast (B) and standard low-fat breakfast (C). Each participant will receive a single oral dose of HMPL-523 acetate tablets 300 mg (3 tablets × 100 mg) on Day 1 of each cycle in accordance with the dosing sequence. During the study, every effort should be made to ensure that the participant takes the medication according to the study protocol.

Administration Method Fasting (A): Participants will fast for at least 10 hours, have blank blood sample collected, and take the study drug with about 240 mL of water. Except for the water for drug administration mentioned above, water will be deprived from 1 hour pre-dose and 1 hour post-dose. Food will be deprived within 4 hours post-dose.

Standard high-fat breakfast (B) or standard low-fat breakfast (C): Participants will fast for at least 10 hours before the standard high-fat breakfast (B) or standard low-fat breakfast (C), start eating breakfast 30 minutes before dosing, and finish the meal within 25 minutes. After the meal, participants will have blank blood sample collected, and take the study drug with about 240 mL of water exactly 30 minutes from the start of the meal. Water will be deprived from 1 hour pre-dose to 1 hour post-dose, except for the beverages included in the prescribed breakfast and water taken with medication. Food will be deprived within 4 hours post-dose.

During hospitalization, the diet of the participants will be provided by the site. On the day of dosing in each cycle, lunch and dinner (both regular meals) will be served 4 hours and 10 hours after dosing, respectively; at other times, 3 meals will be provided according to the schedule arranged by the site.

The dosing period consists of three cycles, and the scheduled PK blood sampling time points for each participant in each cycle are as follows: within 0.5 hours pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60,and 72 hours post-dose, with a total of 18 collections, and about 3 mL of venous blood will be collected each time. The 4-hour post-dose blood sample must be taken prior to lunch.

After the participants are admitted to the clinical study ward, the vital sign measurements will be performed 1 day pre-dose in each cycle and 3±1 hours post-dose on Day 1 of each cycle. Vital sign measurements, blood chemistry, and hematology will be performed on Day 4 of the each of Cycle 1 and Cycle 2. On Cycle 3 Day 4, the participants will be discharged after vital sign measurements, physical examination, laboratory tests, and 12-lead ECG examination are completed.

Strenuous exercise, alcohol, tobacco, tea, and caffeinated beverages should be avoided during the study. Seville oranges, grapefruits or beverages containing these fruits should be avoided during the study.

Follow-up Period Participants will be followed up to Day 12±2 after the last dose (the day of the last dose is defined as Day 1 of follow-up period). The investigator will collect all (adverse events) AEs and concomitant medications/therapies from the participants during this period through telephone calls (or other means such as text messages). If there are AEs ongoing at follow-up, follow-up will continue until the events return to normal level, abnormal and not clinically significant, baseline level, stable or lost to follow-up, or refusal to visit, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Participants can communicate well with the investigator, voluntarily sign the ICF, and agree to comply with the requirements of the study protocol;
2. Male and female healthy participants aged 18-45 years (inclusive);
3. Body weight ≥ 45 kg (females), or ≥ 50 kg (males), body mass index (BMI) 19-26 kg/m2 (inclusive);
4. Participants must commit to using highly effective contraception for both themselves and their sexual partners during the study, and for 180 days after the end of the last study dose, and must not engage in sperm donation, egg donation, or have birth plan.

Exclusion Criteria:

1. Abnormal and clinically significant results of vital signs, physical examination, 12-lead ECG, chest X-ray (frontal and lateral), laboratory tests (including hematology, blood chemistry, urinalysis, etc.) or serum creatinine above the upper limit of normal at screening;
2. Positive for any of the HBsAg, HCV antibody, HIV antibody, or Treponema pallidum antibody;
3. History or current evidence of severe or chronic metabolic/endocrine, hepatic, renal, hematological, pulmonary, immunological, cardiovascular, gastrointestinal, genitourinary, neurological or psychiatric diseases;
4. Prior history of hypertension;
5. Prior history of severe gastrointestinal diseases such as dysphagia, active gastric ulcers, etc., resulting in inability to take oral medication or disorders in absorption of oral medication
6. Prior history of gastrointestinal surgery, renal surgery, cholecystectomy, etc. that, in the judgment of the investigator, may affect drug absorption or excretion;
7. Prior history of drug allergy, or acute allergic rhinitis or food allergy within 2 weeks before screening, or allergy to the active ingredients or excipients of the study drug;
8. Use of any prescription drugs and Chinese herbal medicines within 30 days prior to the first dose;
9. Use of any over-the-counter drugs, vitamins, and health products within 14 days prior to the first dose;
10. Consumption of more than 10 cigarettes per day within 3 months before screening, or those who cannot quit smoking during the study;
11. Regular alcohol consumption within 6 months before screening, that is, those who drink more than 14 units of alcohol per week (1 unit = 360 mL of beer, or 45 mL of spirits with an alcohol content of 40%, or 150 mL of wine), or those who cannot abstain from alcohol during the study, or those who are positive for alcohol breath test;
12. History of drug abuse or recreational use, or positive for urine drug abuse screen;
13. Blood donation (including blood component donation) or blood loss ≥ 400 mL within 3 months prior to screening, use of blood products within 2 months prior to screening, blood donation (including component blood donation) or lost blood ≥ 200 mL within 1 month prior to screening, or a plan to donate blood or blood components during the study or within 1 month after the end of the study;
14. Difficulty in blood collection, or a history of needle phobia or blood phobia, or intolerance to blood sampling via venipuncture, or poor evaluation of venous blood collection;
15. Those who have participated in clinical trials of other drugs/medical devices and have taken study drugs within 3 months prior to screening;
16. Those who have consumed foods, juices or drinks containing alcohol, grapefruit, Seville oranges and caffeine within 72 hours before the first dose, or cannot avoid them during the study;
17. Those who have received live vaccines within 8 weeks prior to screening or have plans to be vaccinated during the clinical trial;
18. Those who have special dietary requirements and cannot accept a standardized dietary arrangement;
19. Pregnant or lactating females, or females with blood pregnancy test results above the upper limit of normal during the screening period, or females with unprotected sex within 2 weeks prior to dosing;
20. The study participant, based on the judgment of the investigator, has any other diseases or conditions that may affect the normal completion of the study or the evaluation of study data, or other conditions that make him/her unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-02-06 (Actual)

PRIMARY OUTCOMES:
AUC0-t | up to one months
  Area under the plasma concentration-time curve from time zero to the last time point t where the concentration could be accurately determined
AUC0-∞ | up to one months
  Area under the plasma concentration-time curve from time 0 to infinity
Cmax | up to one months
  Maximum plasma concentration
Tmax | up to one months
  Other PK parameters of HMPL-523, such as time to Cmax
t1/2 | up to one months
  Other PK parameters of HMPL-523, such as terminal elimination half-life

SECONDARY OUTCOMES:
Adverse events rate | up to one months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Laboratory tests | up to one months
  Number of participants with abnormal laboratory tests results

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Doctor, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No